CLINICAL TRIAL: NCT00367913
Title: Treatment of Pulmonary Disease Caused by MAIS, M.Xenopi or M.Malmoense: A Comparison of Two Triple Drug Regimens and an Assessment of the Value of Immunotherapy With M.Vaccae
Brief Title: Clarithromycin v Ciprofloxacin Added to Rifampicin + Ethambutol, for Opportunist Mycobacterial Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: British Thoracic Society (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BTS Opportunist Mycobacteria
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2006-07

CONDITIONS: Pulmonary Diseases
Keywords: pulmonary disease; Treatment of Opportunist Mycobacteria; Clarithromycin; Ciprofloxacin; M.vaccae; Pulmonary diseases caused by Opportunist Mycobacteria
MeSH Terms: conditions — Lung Diseases | interventions — Ethambutol; Vaccination

INTERVENTIONS:
Drug: Addition of clarithromycin to rifampicin and ethambutol
Drug: Addition of Ciprofloxacin to rifampicin and ethambutol
Biological: Vaccination with M.vaccae

SUMMARY:
To date key drugs in the treatment of MAIS, M.malmoense and M.xenopi (Opportunist Mycobacteria have been rifampicin and ethambutol. Clarithromycin and Ciprofloxacin are active in vitro against these species of mycobacteria. The primary aim of this study was to compare these to agents as supplements to rifampicin and ethambutol. A secondary aim was to assess the vale of immunotherapy with M.vaccae.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary disease due to M.avium intracellulare, M.malmoense or M.xenopi. Aged 16 or over. With clinical and/or radiological evidence of active infection and producing sputum positive on culture on at least 2 occasions.

Exclusion Criteria:

* Pregnant women and women of childbearing age not taking adequate contraceptive precautions.

Patients who have sputum currently positive on culture for M.tuberculosis or M.bovis.

Patients who have AIDS or who are known to be HIV positive

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1995-03; Study Completion 2004-09

PRIMARY OUTCOMES:
Death rates
Cure rates
Relapse rates
Unwanted effects of therapy

SECONDARY OUTCOMES:
Benefit or not of immunotherapy with M.vaccae

CONTACTS AND LOCATIONS:
Overall Officials: Ian Campbell, BSc MD FRCP, Principal Investigator — British Thoracic Society, Research Committee
Locations (1):
- Llandough Hospital, Penarth, Vale of Glamorgan, United Kingdom